CLINICAL TRIAL: NCT00206726
Title: Phase II Study Using Alemtuzumab Combined With Fludarabine for the Treatment of Relapsed/Refractory B-cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Alemtuzumab/Fludarabine for Relapsed/Refractory B-cell Chronic Lymphocytic Leukemia (B-CLL)
Acronym: ECO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13603; 305825 (Other: Sanofi)
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; fludarabine

ARMS (1):
- Alemtuzumab plus Fludarabine (Experimental): Alemtuzumab (Campath) 30mg subcutaneous (SC) plus Fludarabine (Fludara) 25mg/m² intravenous (IV), Days 1-5 every 28 days.
  Interventions: Drug: Alemtuzumab plus Fludarabine

INTERVENTIONS:
Drug: Alemtuzumab plus Fludarabine — Alemtuzumab (Campath) 30mg subcutaneous (SC) plus Fludarabine (Fludara) 25mg/m² intravenous (IV), Days 1-5 every 28 days

SUMMARY:
This is a multi-center, Phase II, open label trial evaluating the efficacy and safety of alemtuzumab and fludarabine in the treatment of B-cell chronic lymphocytic leukemia (B-CLL) patients who have received at least one prior therapy.

Treatments will be administered on a 28-day cycle for 4-6 cycles, with an evaluation during Cycle 4 to permit re-staging. Alemtuzumab and fludarabine will be administered on Days 1-5 of each cycle. Patients will be assessed for response at the time of re-staging at Cycle 4 and at the end of Cycle 6. At the time of the re-staging, patients achieving a Partial Remission (PR) or Stable Disease (SD) will be given an additional 2 cycles of treatment and patients demonstrating presumptive signs of a Complete Remission (CR) will receive no further treatment but will be followed for response.

DETAILED DESCRIPTION:
As of April, 2011 Bayer transferred this record to Genzyme. Genzyme is now the sponsor of this trial. NOTE: This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have confirmed B-CLL.
* Patients must have received at least one prior therapy and must require treatment for active disease

Exclusion Criteria:

* Treatment with any anti-cancer agents (chemotherapies, monoclonal antibodies, etc) within 4 weeks of start of study.
* History of significant allergic reaction to antibody therapies that required discontinuation of antibody therapy
* History of human immunodeficiency virus (HIV) positivity.
* Active infection requiring treatment
* Pregnancy or lactation
* Other severe, concurrent diseases or mental disorders
* Central nervous system involvement of chronic lymphocytic leukemia (CLL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- United States (27):
  - Birmingham, Alabama
  - Berkeley, California
  - Burbank, California
  - Concord, California
  - Stanford, California
  - Washington D.C., District of Columbia
  - Lakeland, Florida
  - Atlanta, Georgia
  - Aurora, Illinois
  - Chicago, Illinois
  - Springfield, Illinois
  - Metairie, Louisiana
  - Clinton, Maryland
  - Boston, Massachusetts
  - Jackson, Michigan
  - Minneapolis, Minnesota
  - Reno, Nevada
  - Lebanon, New Hampshire
  - New Brunswick, New Jersey
  - Albany, New York
  - Northport, New York
  - Lawton, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Johnson City, Tennessee
  - Tacoma, Washington
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in the United States from 12 May 2005 (date of first participant's first visit) to 10 April 2008 (date of last participant's last visit)
Pre-assignment Details: 66 screened, 6 screen failures, 60 enrolled and registered (Intent-to-Treat [ITT] population), 3 withdrew consent prior to receiving therapy = 57 treated (Safety population); 41 received at least 4 therapy cycles with no major protocol deviation or progressed/relapsed or died before completing 4 cycles (Per Protocol [PP] population)
Period: Overall Study
Arm/Group | Alemtuzumab Plus Fludarabine
Started | 60
Treatment Started | 57 (Safety population (3 withdrew consent prior to receiving study drug))
4 Cycles Completed | 41 (per protocol population)
Completed | 9 (4-6 cycles of treatment with assessments at 2, 6, and 9 months post last dose)
Not Completed | 51
Not completed — Delayed recovery of blood counts | 1
Not completed — Progressive disease or relapsed disease | 18
Not completed — Placed on new protocol | 1
Not completed — Bone marrow transplant | 1
Not completed — Adverse Event | 17
Not completed — Death | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Beta 2-micro-globulin [Number; unit: Participants] — Blood serum levels
  Participants
    < 2 milligrams per liter (mg/L) or missing | 12
    >= 2mg/L | 48
Lymph node size [Number; unit: participants] — Bidimensional measurement by palpation
  participants
    < 5 centimeters (cm) | 43
    >= 5 cm | 12
    missing | 5
Number of prior cancer therapies [Number; unit: Participants]
  1 | 10
  2 | 14
  3 | 13
  4 | 5
  5-10 | 16
  >10 | 2
Rai Stage [Number; unit: participants] — Staging system for chronic lymphocytic leukemia (CLL) based on lymphocyte count and percent lymphocytes in bone marrow plus enlarged lymph nodes, or enlarged spleen or liver, or anemia, or thrombocytopenia
  participants
    0 | 5
    1 to 2 | 22
    3 to 4 | 33
    Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: Participants evaluated for therapeutic clinical response according to National Cancer Institute (NCI) response criteria, 28 days after 4 or 6 treatment cycles. Response confirmation involved bone marrow biopsy and aspirate performed 2 months after final treatment. CR requires for at least 2 months: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count (CBC); confirmed by bone marrow aspirate and biopsy 2 months later with lymphocytes <30% of nucleated cells and procedure repeated in 4 weeks if hypocellular.
Time Frame: 28 days after last cycle with confirmation 2 months later
Population: ITT population (all enrolled and registered subjects).
Measure: Number; unit: Percentage of participants with CR
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 60
Percentage of participants with CR | 8.3
Statistical Analysis 1: Comparison: Alemtuzumab Plus Fludarabine; Comparison of CR rate versus 2 percent (%) historic control (p-value and 90% confidence interval); Test type: Superiority or Other; p = 0.014, exact binomial test — 2-sided p-value computed from an exact binomial test comparing the observed rate versus 2% historical rate; CR rate = 0.0833, 90% CI [0.0334 to 0.1673]

2. Secondary Outcome: Overall Response (OR)
Description: Participant had either complete response (CR) or partial response (PR) at 28 days after last treatment cycle (date of OR) and at Months 2 follow-up. PR requires for at least 2 months: 50% decrease from Baseline in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence or absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin, or 50% improvement from Baseline for these parameters without transfusions, nodular CR or persistent anemia/thrombocytopenia unrelated to disease.
Time Frame: 28 days after last cycle with confirmation 2 months later
Population: ITT Population (all subjects enrolled and registered).
Measure: Number; unit: Percentage of participants with CR or PR
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 60
Percentage of participants with CR or PR | 28.3

3. Secondary Outcome: Overall Survival (OS)
Description: Percentage of participants alive 1 year after the first dose date, described as Kaplan-Meier estimate at 1 year
Time Frame: 1 year after start of treatment
Population: Safety Population (all subjects treated)
Measure: Number; unit: Percentage of participants alive
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 57
Percentage of participants alive | 86.4

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Percentage of participants who survived progression-free at 1 year, described as Kaplan-Meier estimate at 1 year
Time Frame: 1 year after start of treatment
Population: ITT population (all subjects enrolled and registered). As three subjects never received study medication, they were to be censored at day 1 for all time-to-event analyses. Thus, the Kaplan-Meier estimates beyond day one are the same for both, the ITT and the safety population.
Measure: Number; unit: percentage alive without progression
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 60
percentage alive without progression | 48.8

5. Secondary Outcome: Percentage of Participants With Overall Response at Different Observation Times
Description: Participant had either complete response (CR) or partial response (PR) at different observation times (after 90 days; after 180 days; after 270 days). PR requires for at least 2 months: 50% decrease from Baseline in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence or absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin, or 50% improvement from Baseline for these parameters without transfusions, nodular CR or persistent anemia/thrombocytopenia unrelated to disease.
Time Frame: from first date of confirmed response until relapse, or death, or study data cutoff date, whichever is earlier
Population: Subjects who achieved Overall Response (OR) defined as number of subjects who achieved CR + number of subjects who achieved PR
Measure: Number; unit: percentage of participants in response
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 17
percentage of participants in response
  After 90 days | 76.5
  After 180 days | 64.7
  After 270 days | 29.4

6. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD)
Description: Presence of MRD was assessed by laboratory testing of molecular responses in blood and bone marrow samples.
Time Frame: When CR is confirmed
Population: All participants for whom CR was confirmed
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Plus Fludarabine
Number analyzed (Participants) | 5
participants
  Positive | 3
  Negative | 2
  Not Assessed | 0

ADVERSE EVENTS:
Arm/Group | Alemtuzumab Plus Fludarabine
Serious Adverse Events (participants affected / at risk) | 41/57
Other Adverse Events (participants affected / at risk) | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab Plus Fludarabine (N=57)
Abdominal pain (Gastrointestinal disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 9
Angina pectoris (Cardiac disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Asthenia (General disorders) | 2
Bacteraemia (Infections and infestations) | 2
Blastomycosis (Infections and infestations) | 1
Blood calcium decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Bronchopneumonia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Chills (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Coagulopathy (Blood and lymphatic system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Disease progression (General disorders) | 3
Disorientation (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Enterococcal bacteriaemia (Infections and infestations) | 1
Epstein-Barr virus test positive (Investigations) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Headache (Nervous system disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxic encephalopathy (Nervous system disorders) | 1
Infection (Infections and infestations) | 1
Influenza like illness (General disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Liver abscess (Infections and infestations) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Multi-organ failure (General disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myelitis (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Obstructive uropathy (Renal and urinary disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Pneumonia (Infections and infestations) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Prolymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 11
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 3
Renal tubular necrosis (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Sepsis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Septic shock (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Sinusitis fungal (Infections and infestations) | 1
Splenic abscess (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab Plus Fludarabine (N=57)
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 30
Anorexia (Metabolism and nutrition disorders) | 13
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate Aminotransferase increased (Investigations) | 3
Asthenia (General disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Axillary pain (General disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bacterial test positive (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 3
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin unconjugated increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Body tinea (Infections and infestations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Breast pain (Reproductive system and breast disorders) | 1
Bronchitis (Infections and infestations) | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Calcium deficiency (Metabolism and nutrition disorders) | 1
Candidiasis (Infections and infestations) | 1
Cardiac murmur (Investigations) | 1
Chapped lips (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 18
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic sinusitis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Confusional state (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 15
Contusion (Injury, poisoning and procedural complications) | 3
Convulsion (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 2
Cytomegalovirus infection (Infections and infestations) | 2
Cytomegalovirus test positive (Investigations) | 22
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 3
Depression (Psychiatric disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 19
Diplopia (Eye disorders) | 1
Disease progression (General disorders) | 13
Disorientation (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 7
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Dysuria (Renal and urinary disorders) | 1
Ear infection (Infections and infestations) | 1
Ear pain (Ear and labyrinth disorders) | 3
Early satiety (General disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Eosinophilia (Blood and lymphatic system disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Face oedema (General disorders) | 1
Facial palsy (Nervous system disorders) | 1
Faeces hard (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 30
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Genital pruritus female (Reproductive system and breast disorders) | 1
Gingival infection (Infections and infestations) | 2
Glossodynia (Gastrointestinal disorders) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Goitre (Endocrine disorders) | 1
Granulocyte count decreased (Investigations) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 6
Haematuria (Renal and urinary disorders) | 1
Haemoglobin decreased (Investigations) | 4
Haemolysis (Blood and lymphatic system disorders) | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Headache (Nervous system disorders) | 6
Heart rate increased (Investigations) | 1
Heart sounds abnormal (Investigations) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hernia pain (General disorders) | 1
Herpes zoster (Infections and infestations) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hot flush (Vascular disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypoaesthesia (Nervous system disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypogammaglobulinaemia (Immune system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 8
Hypothermia (General disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Immunosuppression (Immune system disorders) | 1
Infection (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Injection site erythema (General disorders) | 5
Injection site irritation (General disorders) | 1
Injection site pain (General disorders) | 3
Injection site rash (General disorders) | 1
Injection site reaction (General disorders) | 3
Injection site warmth (General disorders) | 1
Insomnia (Psychiatric disorders) | 7
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 18
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Local swelling (General disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Lymphocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Magnesium deficiency (Metabolism and nutrition disorders) | 1
Medical device pain (Injury, poisoning and procedural complications) | 1
Memory impairment (Nervous system disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Micturition disorder (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Mucosal erosion (General disorders) | 1
Mucosal inflammation (General disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscucoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Mycobacterium avium complex infection (Infections and infestations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 32
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 34
Neutrophil count decreased (Investigations) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 6
Non-cardiac chest pain (General disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 7
Oesophagitis (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pallor (Vascular disorders) | 1
Palpitations (Cardiac disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 3
Pharyngitis (Infections and infestations) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Platelet count decreased (Investigations) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pollakiuria (Renal and urinary disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 27
Rash (Skin and subcutaneous tissue disorders) | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Red blood cell count decreased (Investigations) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Sepsis (Infections and infestations) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Sinus Tachycardia (Cardiac disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus headache (Nervous system disorders) | 1
Sinusitis (Infections and infestations) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Suprapubic pain (General disorders) | 1
Syncope (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 6
Testicular pain (Reproductive system and breast disorders) | 1
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 26
Tinnitus (Ear and labyrinth disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Transaminases increased (Investigations) | 2
Tremor (Nervous system disorders) | 2
Troponin increased (Investigations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Viral DNA test positive (Investigations) | 1
Vision blurred (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 18
Weight decreased (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
White blood cell count decreased (Investigations) | 7
White blood cell disorder (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No